CLINICAL TRIAL: NCT03937596
Title: A Randomized Placebo-controlled Trial of Adjunctive D-cycloserine in Repetitive Transcranial Magnetic Stimulation for Major Depressive Disorder
Brief Title: Adjunctive D-Cycloserine in Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB18-2142
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- D-Cycloserine (Experimental): Participants will orally ingest a capsule containing 100mg of the antibiotic d-cycloserine daily (Monday-Friday) for the first 2 weeks of rTMS treatment (10 sessions), followed by 2 weeks of rTMS without adjunctive medication.
  Interventions: Drug: D-cycloserine; Device: Transcranial Magnetic Stimulator
- Placebo (Placebo Comparator): Participants will orally ingest a capsule identical to that containing the study medication, however this capsule will contain a placebo. They will ingest this capsule daily (Monday-Friday) for the first 2 weeks of rTMS treatment (10 sessions), followed by 2 weeks of rTMS without adjunctive medication.
  Interventions: Device: Transcranial Magnetic Stimulator; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: D-cycloserine — Daily oral D-cycloserine 100mg during the blinded phase (10 days).
  Other Names: Seromycin
  Arms: D-Cycloserine
Device: Transcranial Magnetic Stimulator — Repetitive Transcranial magnetic stimulation (rTMS) will be delivered using a MagPro X100 device with B70 coil and the intermittent theta burst (iTBS) protocol to the left dorsolateral prefrontal cortex. Participants will receive daily treatments (Monday-Friday) over four weeks.
Drug: Placebo oral capsule — Daily oral placebo during the blinded phase (10 days).
  Arms: Placebo

SUMMARY:
Transcranial magnetic stimulation (rTMS) is an approved treatment for depression. The purpose of this study is to test an adjunctive medication, D-cycloserine, in rTMS for depression using a placebo-controlled design. D-Cycloserine is a partial N-Methyl-D-Aspartate receptor (NMDAr) agonist, and therefore may enhance the effects of rTMS, however there is data to support and refute this hypothesis. Using a double-blind design, the investigators will randomize patients with Major Depressive Disorder to receive either daily low dose D-cycloserine or placebo in conjunction with rTMS to the left dorsolateral prefrontal cortex. After 10 treatments (2 weeks), this double-blind period will conclude and all participants will receive an additional 10 treatments (2 weeks) of rTMS without any adjuncts. The primary outcome will be improvement in clinician rated depressive symptoms at the conclusion of the study.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a common and debilitating illness. For an unacceptable proportion of patients, depressive symptoms remain impairing despite multiple treatments. Increasingly, non-invasive brain stimulation techniques are being explored as a means of targeting specific brain regions and networks that are implicated in depression. Repetitive transcranial magnetic stimulation (rTMS) is the non-invasive stimulation technique with the largest evidence base in MDD. Targeting the dorsolateral prefrontal cortex (DLPFC) with rTMS has proven an effective treatment for MDD, however as many as 2/3 of patients will not experience substantial improvement. Adjunctive agents are a potential strategy to improve patient outcomes.

The objective of the proposed study is to determine the efficacy of adjunctive D-cycloserine with rTMS directed to the left dorsolateral prefrontal cortex (DLPFC) in acute Major Depressive Episodes. The investigators propose to utilize a stimulation protocol called the intermittent theta-burst protocol to study rTMS in conjunction with D-cyloserine using a randomized double-blind, placebo-controlled design with allocation concealment. Patients with Major Depressive Disorder will be randomized to receive 1) rTMS+cycloserine, or 2) rTMS+placebo in a 1:1 ratio for two weeks (10 sessions).

At the conclusion of the 2-week blinded augmentation phase, patients will continue to receive two weeks of rTMS without an augmentation agent or placebo.

The primary outcome measures will be improvement in depression as measured by change in Montgomery Asberg Depression Rating Scale (MADRS). In addition, the investigators will also be looking at the improvement of other clinical outcome measures, quality of life and changes in brain functional dynamics, as assessed with functional Magnetic Resonance Imaging (MRI), and metabolites, as assessed by Magnetic Resonance (MR) Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* are competent to consent to treatment
* have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of DSM-5 criteria Major Depressive Disorder with a current episode of at least moderate severity of depression, single or recurrent
* have failed to achieve a clinical response to one adequate trial of antidepressant medication within the current episode, or been unable to tolerate antidepressant medications.
* have a score ≥ 18 on the Hamilton Depression Rating Scale 17-item
* have a Young Mania Rating Scale Score of ≤ 8
* have had no change in dose, or initiation of any psychotropic medication in the 4 weeks prior to randomization
* are able to adhere to the treatment schedule
* pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria:

* Allergy to Cycloserine
* Have failed adequate trials of ≥4 antidepressant treatments in the current episode.
* have an alcohol or substance use disorder within the last 3 months
* have suicidal ideation (score of 4 ≥ on item 10 of MADRS)
* are at a significant risk of harm to themselves or others
* history of psychosis
* are currently pregnant , breast feeding or plan to become pregnant
* have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of other primary psychiatric diagnoses as assessed by a study investigator to be primary and causing greater impairment than Major Depressive Disorder.
* have failed a course of electroconvulsive therapy (ECT) in the current episode. Previous ECT treatment outside of the current episode does not influence inclusion.
* history of non-response to rTMS treatment.
* have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
* have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
* have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
* are currently (or in the last 4 weeks) taking lorazepam or any other benzodiazepine due to the potential to limit rTMS efficacy
* have an exclusion criteria for MRI: Those with a history of cranial, thoracic or abdominal surgery, with pacemakers, artificial joints or other metallic implants will be excluded from the MRI scan. Subjects that have agreed to participate in the MRI portion of the study will be pre-screened for any potential metal fragments in the body (particularly in the orbits) if they have had any history of doing metal work or have been involved in use/deployment of ammunitions/explosives, welding, piping etc).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Change in severity of depressive symptoms as measured by the MADRS, a clinician-rated instrument. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes. The overall score ranges from 0 - 60. Cutoff points are 0-6 = normal, 7-9 = mild depression, 20-34 = moderate depression, >34 = severe depression.

SECONDARY OUTCOMES:
Functional Magnetic Resonance Imaging (fMRI) | Administered at baseline and week 2. Change in cycloserine group vs change in placebo group
  Change in task and resting state functional connectivity as determined by an fMRI.
Magnetic Resonance (MR) spectroscopy | Administered at baseline and week 2. Change in cycloserine group vs change in placebo group
  Change in brain metabolites in regions of interest.
Clinical Remission | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Score of </= 10 on the MADRS
Clinical Response | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  >/= 50% reduction in MADRS scores
Quality of Life as measured by the World Health Organization Quality of Life (WHOQOL-BREF) questionnaire | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  The WHOQOL-BREF is a self-reported questionnaire which assesses individual's perception of their quality of life across 4 domains; physical health, psychological, social relationships and environment. Domains scores are calculated to range from 0-20 and scaled in a positive direction (ie. higher scores denote higher quality of life).
Anxiety Symptoms | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  Anxiety symptoms will be assessed using the 7 item Generalized Anxiety Disorder (GAD-7) questionnaire. The GAD-7 measures self-reported feelings of anxiety within the last 2 weeks. Scores range from 0-21. Scores of 5, 10, and 15 represent cut points for mild, moderate, and severe anxiety, respectively.
Workplace Productivity | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  Productivity will be assessed using the Lam Employment Absence and Disability Scale (LEAPS). The LEAPS is a 10-item, self-rated scale and provides information on how participants are functioning at work. Scores range from 0 - 28, with higher scores representing more severe work impairment.
Functional Disability | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  Functional disability will be assessed using the Sheehan Disability Scale (SDS). The SDS is a self-report scale to assess functional impairment in three domains; work/school, social and family life. Scores range from 0 - 30, with higher scores representing greater impairment.
Clinical Global Impression | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  Clinical Global Impression will be assessed using the Clinical Global Impression (CGI) Severity and Improvement scales. The CGI-Severity scale is clinician rated from 1-7 representing 'Not at all ill' to 'Severely ill'. The CGI-Improvement scale is also rated 1-7, representing the range between 'Very much improved' and 'Very much worse'.
Cognitive Function | Administered at baseline and at the halfway point (week 2)
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes 4 objective cognitive tests (adapted from choice reaction time, 1-back working memory task, symbol digit coding, and Trails-B) and a subjective cognitive questionnaire (PDQ-5). Results indicate cognitive performance compared to healthy age-, sex- and education-matched individuals.
Implicit Suicidal Thoughts | Administered at baseline and at the halfway point (week 2)
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings
Personality Measures- BFI | Administered at baseline and after rTMS treatment (week 4)
  The Big Five Inventory (BFI) is a self-report inventory designed to measure the Big Five dimensions of personality: extroversion, agreeableness, openness, conscientiousness, and neuroticism. The test consists of 44 items that you must rate on how true they are about you on a five point scale where 1=Disagree, 3=Neutral and 5=Agree.
Personality Measures- DEQ | Administered at baseline and after rTMS treatment (week 4)
  The Depressive Experiences Questionnaire (DEQ) is a 66 item questionnaire where participants rate themselves on life experiences and personality characteristics frequently associated with depression. Participants are asked to rate each item on a seven-point Likert-type scale ranging from strongly disagree (1) to strongly agree (7). Analysis of results produces 3 factors: Dependency, Self-criticism, and Efficacy.
Anhedonia | Administered at baseline and after rTMS treatment (week 4)
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item self report developed to measure ability to experience pleasure (hedonic tone) and its absence (anhedonia) in the last few days. Each item asks participants to agree or disagree with how pleasurable a certain scenario would be. Disagree responses receive a score of 1 and Agree responses receive a score of 0. The SHAPS is scored as the sum of the 14 items so that total scores ranged from 0 to 14. A higher total SHAPS score indicated higher levels of anhedonia.
Self-reported Cognition | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  The Cognitive Failures Questionnaire (CFQ) measures self-reported failures in perception, memory, and motor function in the completion of everyday tasks. Individuals are asked to rate the frequency experiences and behaviors on a 5-point scale: 0-Never, 1-Very rarely, 2-Occasionally, 3-Quite often, 4-Very often.
Depressive Symptoms | Administered at baseline, week 1, at the halfway point (week 2), week 3, and after rTMS treatment (week 4)
  The Quick Inventory of Depressive Symptomatology- Self Report (QIDS-SR) is a scale of self-report measure of depression. Questions in the QIDS - SRcorrelate with the nine DSM-IV symptom criterion domains, Including: Sleep disturbance, Sad mood, Decrease/increase in appetite/weight, Concentration, Self-criticism, Suicidal ideation, Interest, Energy/fatigue, Psychomotor agitation/retardation.Severity of depression can be judged based on the total score.
  1-5 = No depression 6-10 = Mild depression 11-15 = Moderate depression 16-20 = Severe depression 21-27 = Very severe depression
VAS for General Health | Administered at baseline, at the halfway point (week 2), and after rTMS treatment (week 4)
  A Visual Analog Scale (VAS) will ask participants how good or bad their health is today. This scale is numbered from 0 to 100. 100 indicates the best health they can imagine. 0 indicates the worst health they can imagine.
Perception of Illness | Administered at baseline and after rTMS treatment (week 4)
  The Brief Illness Perception Questionnaire (BIPQ) is a nine-item scale designed to rapidly assess the cognitive and emotional representations of illness. The BIPQ assesses perception on a 0 (minimum) -10 (maximum) response scale. It includes 5 items on cognitive representation of illness perception, 2 items on emotional representation, 1 item on illness comprehensibility, and 1 item on perceived cause of illness.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Daily Monday-Friday throughout study (4 weeks)
  Adverse events will be tracked and recorded
Side Effects | Daily Monday-Friday throughout study (4 weeks)
  Side effects will be tracked through a comfort rating questionnaire. The comfort rating questionnaire assesses the frequency and severity of side effects common to rTMS treatment. Severity of side effects are rated from 1 (none) to 10 (extreme).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cole J, Sohn MN, Harris AD, Bray SL, Patten SB, McGirr A. Efficacy of Adjunctive D-Cycloserine to Intermittent Theta-Burst Stimulation for Major Depressive Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2022 Dec 1;79(12):1153-1161. doi: 10.1001/jamapsychiatry.2022.3255. PMID 36223114